CLINICAL TRIAL: NCT03172598
Title: A Phase IIa, Multi-Centre, Randomised, Double-Blind, Cross-Over, Placebo-Controlled Study to Assess the Efficacy, Safety and Tolerability of MT-8554 in Subjects With Painful Diabetic Peripheral Neuropathy Incorporating an Open Label Pilot Arm
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of MT- 8554 in Subjects With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MT-8554-E06
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Painful Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MT-8554 low dose (Experimental): Patients who meet eligibility criteria will be administered twice daily low dose of MT-8554 during the treatment period.
  Interventions: Drug: MT-8554 low dose
- MT-8554 middle dose (Experimental): Patients who meet eligibility criteria will be administered twice daily middle dose of MT-8554 during the treatment period.
  Interventions: Drug: MT-8554 middle dose
- MT-8554 high dose (Experimental): Patients who meet eligibility criteria will be administered twice daily high dose of MT-8554 during the treatment period.
  Interventions: Drug: MT-8554 high dose
- MT-8554, then placebo (Experimental): The study participants will receive MT-8554 (TBD mg) in the first phase, followed by placebo in the second phase
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 middle dose; Drug: MT-8554 high dose; Drug: Placebo
- Placebo, then MT-8554 (Experimental): The study participants will receive placebo in the first phase, followed by MT-8554 (TBD mg) in the second phase
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 middle dose; Drug: MT-8554 high dose; Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 low dose — Capsule
  Arms: MT-8554 low dose; MT-8554, then placebo; Placebo, then MT-8554
Drug: MT-8554 middle dose — Capsule
  Arms: MT-8554 middle dose; MT-8554, then placebo; Placebo, then MT-8554
Drug: MT-8554 high dose — Capsule
  Arms: MT-8554 high dose; MT-8554, then placebo; Placebo, then MT-8554
Drug: Placebo — Capsule
  Arms: MT-8554, then placebo; Placebo, then MT-8554

SUMMARY:
A Study to Investigate the Safety, Tolerability and Efficacy of Multiple Doses of MT-8554 in Subjects with Painful Diabetic Peripheral Neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and female subjects aged ≥18 years
* Subjects who have a history of pain at least 6 months and ≤7 years attributed to diabetic peripheral neuropathy
* A body mass index ranging from 18 to 45 kg/m2

Exclusion Criteria:

* Subjects who have participated in a clinical study of any IMP (other than placebo) within 12 weeks (from last administration) prior to screening or who are currently participation in another clinical study
* Unstable or uncontrolled diabetes
* Clinically significant 12-lead ECG abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by vital signs and Adverse Events | Up to Day 22
  Number of participants with potentially clinically important vital sign measurements or tolerability issues
Efficacy as measured by reduction in pain using a numerical rating scale. | Up to Day 49
  Pain reduction using an 11-point numerical rating scale

SECONDARY OUTCOMES:
Number of subjects with electrocardiogram (ECG) findings of potential clinical importance | Up to Day 49
  Number of participants with potentially clinically important ECG findings
Plasma concentration of MT-8554 | Up to Day 49
  Maximum Observed Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Europe Ltd
Locations (3):
- Investigational center, City Name, Germany
- Investigational center, City Name, Hungary
- Investigational center, City Name, Poland